CLINICAL TRIAL: NCT02851316
Title: The Effect of Whole Body Vibration on Running Biomechanics in Individuals With Anterior Cruciate Ligament Reconstruction
Brief Title: Whole Body Vibration on Running Biomechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Fullerton (Other)
Responsible Party: Principal Investigator, Derek Pamukoff, Assistant Professor, California State University, Fullerton
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CSUFullerton
Record Dates: First submitted 2016-07-19; First posted 2016-08-01 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole Body Vibration (Experimental): The WBV intervention consists of 6 bouts of 60 seconds vibration with 2 minutes of rest in between (30Hz, 2g acceleration) while participants stand on a vibrating platform with their knees bent.
  Interventions: Other: Whole Body Vibration
- Control (No Intervention): The control intervention consists of 6 bouts of 60 seconds with 2 minutes of rest in between while participants stand with their knees bent (no vibration applied).

INTERVENTIONS:
Other: Whole Body Vibration — Participants will stand in a squatted position on a platform that provides a brief vibratory stimuli.
  Arms: Whole Body Vibration

SUMMARY:
Whole body vibration (WBV) acutely improves quadriceps strength, and may improve long-term outcomes in individuals with anterior cruciate ligament reconstruction (ACLR). However, it is unclear if WBV influences athletic tasks such as running. The purpose of this study is to evaluate the influence of WBV on running biomechanics in individuals with ACLR.

DETAILED DESCRIPTION:
Individuals with anterior cruciate ligament reconstruction (ACLR) have deficits in quadriceps muscles function that influences walking and running biomechanics. In the long term, alterations in walking and running contribute to physical disability and the development of knee osteoarthritis. Unfortunately, rehabilitation for the quadriceps muscles is often ineffective, and novel strategies to improve rehabilitation efforts are needed. Whole body vibration (WBV) acutely improves quadriceps strength, and may improve long-term outcomes in individuals with ACLR. However, it is unclear if WBV influences athletic tasks such as running.

Specific Aim 1: The purpose of this study is to determine the effect of WBV on running biomechanics in individuals with ACLR. The investigators hypothesize that WBV will improve running characteristics associated with knee osteoarthritis development.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years
* Unilateral ACL reconstruction
* At least 6 months post-reconstruction
* Recreationally active (at least 20 minutes of physical activity 3 times per week)

Exclusion Criteria:

* History of ACL graft rupture or revision surgery
* Neurological disorder
* Other lower extremity within the 6 months prior to participation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in ground reaction force | Day 1, Prior to and immediately following vibration intervention in a single session (i.e. - acute effects)
  Ground reaction force during running gait
Change in ground reaction force loading rate | Day 1, Prior to and immediately following vibration intervention in a single session (i.e. acute effects)
  Ground reaction force loading rate during running gait
Change in knee flexion excursion | Day 1, Prior to and immediately following vibration intervention in a single session (i.e. acute effects)
  Knee flexion excursion during running gait

CONTACTS AND LOCATIONS:
Overall Officials: Derek N Pamukoff, PhD, Principal Investigator — California State University, Fullerton
Locations (1):
- CSU Fullerton: Biomechanics Laboratory (KHS 021), Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pamukoff DN, Montgomery MM, Choe KH, Moffit TJ, Vakula MN. Effect of Whole-Body Vibration on Sagittal Plane Running Mechanics in Individuals With Anterior Cruciate Ligament Reconstruction: A Randomized Crossover Trial. Arch Phys Med Rehabil. 2018 May;99(5):973-980. doi: 10.1016/j.apmr.2017.11.019. Epub 2018 Jan 31. PMID 29407520